CLINICAL TRIAL: NCT01472848
Title: A Randomized, Double-Blind, Outpatient, Placebo-Controlled, Dose Titration Study Of Gastrointestinal Tolerability Of Pf 05212389 (Oap-189) In Obese Subjects
Brief Title: A Study Of Gastrointestinal Tolerability Of PF05212389 In Obese Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2201010
Record Dates: First submitted 2011-03-14; First posted 2011-11-17 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental)
  Interventions: Drug: PF 05212389 or placebo
- Cohort 2 (Experimental)
  Interventions: Drug: PF 05212389 or placebo
- Cohort 3 (Experimental)
  Interventions: Drug: PF 05212389 or placebo
- Cohort 4 (Experimental)
  Interventions: Drug: PF 05212389 or placebo
- Cohort 5 (Experimental)
  Interventions: Drug: PF 05212389 or placebo
- Cohort 6 (Active Comparator)
  Interventions: Drug: PF 05212389 or placebo

INTERVENTIONS:
Drug: PF 05212389 or placebo — QD SC administration of PF 05212389 (12 subjects) or matching placebo (3 subjects); doses ranging from low to high dose.
  Arms: Cohort 1
Drug: PF 05212389 or placebo — QD SC administration of PF 05212389 (12 subjects) or matching placebo (3 subjects); doses ranging from low to high dose.
  Arms: Cohort 2
Drug: PF 05212389 or placebo — QD SC administration of PF 05212389 (12 subjects) or matching placebo (3 subjects); doses to be determined from the results of previous cohorts
  Arms: Cohort 3
Drug: PF 05212389 or placebo — QD SC administration of PF 05212389 (12 subjects) or matching placebo (3 subjects); doses to be determined from the results of previous cohorts
  Arms: Cohort 4
Drug: PF 05212389 or placebo — QD SC administration of PF 05212389 (12 subjects) or matching placebo (3 subjects); doses to be determined from the results of previous cohorts
  Arms: Cohort 5
Drug: PF 05212389 or placebo — QD SC administration of PF 05212389 (12 subjects) or matching placebo (3 subjects); doses to be determined from the results of previous cohorts
  Arms: Cohort 6

SUMMARY:
This study examines whether a gradual increase of dose improves the gastrointestinal tolerability (nausea and vomiting) of PF05212389

ELIGIBILITY:
Inclusion Criteria:

Obesity

Exclusion Criteria:

Diabetes mellitus (type 1 or type 2) Heart failure Eating disorders Psychiatric disorders History of suicide attempt History of pancreatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
- Incidence, severity and duration of nausea and vomiting collected as adverse events. | Day 1 to day 28

SECONDARY OUTCOMES:
- Change in body weight from baseline | Day 1 to day 28
- Changes in heart rate, systolic and diastolic blood pressure, and ECG parameters from baseline | Day 1 to day 28
- Multiple dose PK parameters of PF 05212389 | Day 1 to day 28
- Treatment modification defined as a decrease in any dose of, or discontinuation from, study medication for any reason | Day 1 to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2201010&StudyName=A%20Study%20Of%20Gastrointestinal%20Tolerability%20Of%20PF05212389%20In%20Obese%20Subjects